CLINICAL TRIAL: NCT05137509
Title: YKL -40 as Anew Biomarker in COVID -19 Patients
Brief Title: YKL -40 as New Biomarker in COVID -19 Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Norhan mostafa Mohamed Abdelal, principle investigator, Assiut University
Other Study IDs: AHGNH
Record Dates: First submitted 2021-11-25; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients Infected by severe acute respiratory syndrome coronavirus 2 (SARS-cov-2): Patients Infected by COVID -19 diagnosed by Reverse transcriptase polymerase chain reaction and computerized tomography
  Interventions: Device: Computerized Tomography
- patients suffering from chronic lung disease: Diagnosed by clinical manifestation and Computerized tomogarphy
  Interventions: Device: Computerized Tomography
- Healthy Individuals: They must be without prior history of chronic inflammation in the lung

INTERVENTIONS:
Device: Computerized Tomography — Using Computerized Tomography for diagnosis COVID -19 patients
  Groups: Patients Infected by severe acute respiratory syndrome coronavirus 2 (SARS-cov-2); patients suffering from chronic lung disease

SUMMARY:
The coronavirus disease-2019 (COVID-19)is a pandemic disease caused by SARS -COV-2 which belongs to the β-coronavirus family . The majority of affected individuals exhibit no or mild to moderate symptoms, but up to 15% of patients develop severe pneumonia with approximately 6% progressing to acute respiratory distress syndrome and multiorgan failure.

Biomarkers are needed to identify patients will suffer rapid disease progression to severe complications and death. Preliminary studies describe vasculitic processes underlying organ damage in seriously ill patients, induced by the activation of inflammatory cascades, complement activation and pro-inflammatory cytokines (i.e. interleukin).

The severity of Vasculitic damage is unfortunately not easily predictable through currently used laboratory biomarkers such as D-dimer or prothrombin time/activated partial thromboplastin time.

The severity of the disease is mainly driven by diffuse interstitial lung diseases. YKL-40 has a pro mitogenic action on pulmonary fibroblasts, increases the activity of macrophages and is associated with inflammatory disorders. In ILD, YKL-40 has been described to be associated with the severity of lung diseases and with the risk of death.

YKL-40 serum levels could therefore be of interest for diagnosis and prognosis since it is at the cross-link between vascular and epithelial lung damage.

.

ELIGIBILITY:
Inclusion Criteria:

* • Group one should be diagnosed by RT-PCR (reverse transcriptase polymerase chain reaction).

  * Healthy individual must be without a prior history of chronic inflammation in the lung.

Exclusion Criteria:

* Patients with acute renal failure (ARF) or multiple organ damage (MOF).

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients come to Assiut university with clinical manifestation of COVID -19
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-30 (Estimated); Primary Completion 2024-10-10 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Using YKL -40 to help in diagnosis of COVID -19 and assessment of disease severity | 2 years
  * 1- To highlight the role of YKL-40 biomarker in diagnosis of COVID -19 and assessment of disease severity.
  * 2- To compare the sensitivity and the specificity of YKL- 40 in relation to other biomarkers used in diagnosis of Covid-19.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chan JF, To KK, Tse H, Jin DY, Yuen KY. Interspecies transmission and emergence of novel viruses: lessons from bats and birds. Trends Microbiol. 2013 Oct;21(10):544-55. doi: 10.1016/j.tim.2013.05.005. Epub 2013 Jun 14. PMID 23770275
- [Result] Chan JF, Kok KH, Zhu Z, Chu H, To KK, Yuan S, Yuen KY. Genomic characterization of the 2019 novel human-pathogenic coronavirus isolated from a patient with atypical pneumonia after visiting Wuhan. Emerg Microbes Infect. 2020 Jan 28;9(1):221-236. doi: 10.1080/22221751.2020.1719902. eCollection 2020. PMID 31987001
- [Result] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Result] Inoue Y, Kaner RJ, Guiot J, Maher TM, Tomassetti S, Moiseev S, Kuwana M, Brown KK. Diagnostic and Prognostic Biomarkers for Chronic Fibrosing Interstitial Lung Diseases With a Progressive Phenotype. Chest. 2020 Aug;158(2):646-659. doi: 10.1016/j.chest.2020.03.037. Epub 2020 Apr 5. PMID 32268131
- [Result] Korthagen NM, van Moorsel CH, Barlo NP, Ruven HJ, Kruit A, Heron M, van den Bosch JM, Grutters JC. Serum and BALF YKL-40 levels are predictors of survival in idiopathic pulmonary fibrosis. Respir Med. 2011 Jan;105(1):106-13. doi: 10.1016/j.rmed.2010.09.012. PMID 20888745
- [Result] Lei J, Kusov Y, Hilgenfeld R. Nsp3 of coronaviruses: Structures and functions of a large multi-domain protein. Antiviral Res. 2018 Jan;149:58-74. doi: 10.1016/j.antiviral.2017.11.001. Epub 2017 Nov 8. PMID 29128390
- [Result] Zhang XZ. [CT investigation of spinal injury]. Zhonghua Fang She Xue Za Zhi. 1988 Aug;22(4):227-30. No abstract available. Chinese. PMID 3208584